CLINICAL TRIAL: NCT03925896
Title: LMP2 Antigen-specific High-affinity T Cell Receptor (TCR)-Transduced Autologous T-cell Therapy for Recurrent and Metastatic Nasopharyngeal Carcinoma, an Open-label, Single-center, Phase I Clinical Trial
Brief Title: Phase I Trial of LMP2 Antigen-specific TCR T-cell Therapy for Recurrent and Metastatic NPC Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, MD,PhD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-021
Record Dates: First submitted 2019-04-20; First posted 2019-04-24 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: EBV TCR-T cells; recurrent; metastatic
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LMP2 Antigen-specific TCR T cells (Experimental): All enrolled subjects will be infused with EBV TCR-T cells. The project which enrolls 27 patients, according to the patient's HLA subtypes will be divided into HLA-A2, HLA-A11, HLA-A24 three groups, 9 patients in each group. Using a dose climbing method, each group will be divided into three dose subgroups. In the first dose subgroup, 5×106/kg TCR-T cells will be returned, and in the second dose subgroup, 1×107/kg TCR-T cells will be returned. The third dose subgroup 5 x 107/kg TCR-T cells will be returned.
  Interventions: Drug: LMP2 Antigen-specific TCR T cells

INTERVENTIONS:
Drug: LMP2 Antigen-specific TCR T cells — All enrolled subjects will be infused with EBV TCR-T cells. The project which enrolls 27 patients, according to the patient's HLA subtypes will be divided into HLA-A2, HLA-A11, HLA-A24 three groups, 9 patients in each group. Using a dose climbing method, each group will be divided into three dose subgroups. In the first dose subgroup, 5×106/kg TCR-T cells will be returned, and in the second dose subgroup, 1×107/kg TCR-T cells will be returned. The third dose subgroup 5 x 107/kg TCR-T cells will be returned.
  Other Names: EBV specific TCR-T cells

SUMMARY:
In this study, a single-arm, open-labeled clinical trial will be performed to determine the safety and efficacy of EBV TCR-T cells in the treatment of recurrent/metastatic nasopharyngeal carcinoma with positive EBV infection in the Chinese population.

DETAILED DESCRIPTION:
All enrolled subjects will be infused with EBV TCR-T cells. The project which enrolls 27 patients, according to the patient's HLA subtypes will be divided into HLA-A2, HLA-A11, HLA-A24 three groups, 9 patients in each group. Using a dose climbing method, each group will be divided into three dose subgroups. In the first dose subgroup, 5×106/kg TCR-T cells will be returned, and in the second dose subgroup, 1×107/kg TCR-T cells will be returned. The third dose subgroup 5 x 107/kg TCR-T cells will be returned.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with nasopharyngeal carcinoma diagnosed by pathology and EBV infection (EBERs positive ) ; 2.18-70 years old; 3.MHC-I is HLA-A2, HLA-A11 or HLA-A24 subtype; 4. Progression after second-line platinum-containing chemotherapy regimen, recurrent/metastatic nasopharyngeal carcinoma patients who are inoperable and non-radiable; 5. Based on the Response Evaluation Criteria in Solid Tumors version (RECIST 1.1), there are ≥ 1 measurable target lesions; 6. Expected survival time is more than 12 weeks; 7. ECOG score 0-2 points; 8. Patients with good bone marrow, kidney, liver, and heart, and lung function 9. Can establish the venous access required for the collection, no contraindications for white blood cell collection; 10. Male and female patients of the appropriate age must adopt a reliable method of contraception; 11. Those who understand the trial and have signed an informed consent form.

Exclusion Criteria:

1. Patients with symptomatic brain metastasis;
2. Other malignant tumors other than nasopharyngeal carcinoma within 5 years prior to enrollment, in addition to appropriate treatment of cervical carcinoma in situ, cutaneous basal or squamous cell carcinoma, localized prostate cancer or ductal carcinoma in situ after radical surgery ;
3. Hepatitis B or hepatitis C active period, HIV-infected;
4. Any other uncontrolled active disease that impedes participation in the trial;
5. Patients with severe heart and cerebrovascular diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, and cerebral hemorrhage;
6. 2-3 grade hypertension or patients with poorly controlled hypertension;
7. Those with a history of mental illness that are difficult to control;
8. The investigator believes that it is not appropriate to participate in the trial;
9. Those who have been using immunosuppressive agents for a long time after organ transplantation, except for recent or current inhaled corticosteroids;
10. In the opinion of the investigator, the presence of medical history or mental state history or laboratory abnormalities may increase the risk associated with participating in the study or study drug administration, or may interfere with the interpretation of the results;
11. Screening indicates that the target cell transfection rate is less than 30%, or the T cell expansion is insufficient (less than 5 times) under CD3/CD28 stimulation conditions;
12. Unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events occurred 30 days or 30 days prior to grouping. If receiving anticoagulant therapy, the subject's therapeutic dose must be stable before grouping;
13. A subject who is pregnant or breastfeeding, or who is planning a pregnancy during or after 2 months of treatment;
14. Subjects who are women of childbearing age who are reluctant to receive high-efficiency contraception (according to institutional standards) during treatment and at least 2 months after the end of treatment. Female subjects of childbearing age are required to provide a negative result of a serum or urine pregnancy test within 48 hours prior to treatment;
15. There are active or uncontrollable infections requiring systemic treatment within 14 or 14 days prior to grouping;
16. Subjects who are unwilling or unable to comply with the research requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
To Determine the Maximum Tolerated Dose of TCR T-cell Therapy | 2 years
  Verify the MTD of LMP2 Antigen-specific TCR T-cell Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hai Qiang Mai, MD,PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao WH, Yang LF, Liu XY, Zhou GF, Jiang WZ, Hou BL, Sun LQ, Cao Y, Wang XY. DCE-MRI assessment of the effect of Epstein-Barr virus-encoded latent membrane protein-1 targeted DNAzyme on tumor vasculature in patients with nasopharyngeal carcinomas. BMC Cancer. 2014 Nov 18;14:835. doi: 10.1186/1471-2407-14-835. PMID 25407966
- [Background] Rosenberg SA, Packard BS, Aebersold PM, Solomon D, Topalian SL, Toy ST, Simon P, Lotze MT, Yang JC, Seipp CA, et al. Use of tumor-infiltrating lymphocytes and interleukin-2 in the immunotherapy of patients with metastatic melanoma. A preliminary report. N Engl J Med. 1988 Dec 22;319(25):1676-80. doi: 10.1056/NEJM198812223192527. PMID 3264384
- [Background] Huang J, Fogg M, Wirth LJ, Daley H, Ritz J, Posner MR, Wang FC, Lorch JH. Epstein-Barr virus-specific adoptive immunotherapy for recurrent, metastatic nasopharyngeal carcinoma. Cancer. 2017 Jul 15;123(14):2642-2650. doi: 10.1002/cncr.30541. Epub 2017 Feb 21. PMID 28222215
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Morgan RA, Dudley ME, Wunderlich JR, Hughes MS, Yang JC, Sherry RM, Royal RE, Topalian SL, Kammula US, Restifo NP, Zheng Z, Nahvi A, de Vries CR, Rogers-Freezer LJ, Mavroukakis SA, Rosenberg SA. Cancer regression in patients after transfer of genetically engineered lymphocytes. Science. 2006 Oct 6;314(5796):126-9. doi: 10.1126/science.1129003. Epub 2006 Aug 31. PMID 16946036
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- [Background] Kobayashi E, Mizukoshi E, Kishi H, Ozawa T, Hamana H, Nagai T, Nakagawa H, Jin A, Kaneko S, Muraguchi A. A new cloning and expression system yields and validates TCRs from blood lymphocytes of patients with cancer within 10 days. Nat Med. 2013 Nov;19(11):1542-6. doi: 10.1038/nm.3358. Epub 2013 Oct 13. PMID 24121927
- [Background] Khalil DN, Smith EL, Brentjens RJ, Wolchok JD. The future of cancer treatment: immunomodulation, CARs and combination immunotherapy. Nat Rev Clin Oncol. 2016 May;13(5):273-90. doi: 10.1038/nrclinonc.2016.25. Epub 2016 Mar 15. PMID 26977780
- [Background] Kalos M, Levine BL, Porter DL, Katz S, Grupp SA, Bagg A, June CH. T cells with chimeric antigen receptors have potent antitumor effects and can establish memory in patients with advanced leukemia. Sci Transl Med. 2011 Aug 10;3(95):95ra73. doi: 10.1126/scitranslmed.3002842. PMID 21832238
- [Background] Jackson HJ, Rafiq S, Brentjens RJ. Driving CAR T-cells forward. Nat Rev Clin Oncol. 2016 Jun;13(6):370-83. doi: 10.1038/nrclinonc.2016.36. Epub 2016 Mar 22. PMID 27000958
- [Background] Mueller KT, Maude SL, Porter DL, Frey N, Wood P, Han X, Waldron E, Chakraborty A, Awasthi R, Levine BL, Melenhorst JJ, Grupp SA, June CH, Lacey SF. Cellular kinetics of CTL019 in relapsed/refractory B-cell acute lymphoblastic leukemia and chronic lymphocytic leukemia. Blood. 2017 Nov 23;130(21):2317-2325. doi: 10.1182/blood-2017-06-786129. Epub 2017 Sep 21. PMID 28935694
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Draper LM, Kwong ML, Gros A, Stevanovic S, Tran E, Kerkar S, Raffeld M, Rosenberg SA, Hinrichs CS. Targeting of HPV-16+ Epithelial Cancer Cells by TCR Gene Engineered T Cells Directed against E6. Clin Cancer Res. 2015 Oct 1;21(19):4431-9. doi: 10.1158/1078-0432.CCR-14-3341. PMID 26429982